CLINICAL TRIAL: NCT06100549
Title: Feasibility of Using National Bowel Screening Programme Surplus qFIT Samples to Investigate the Gut Microbiota.
Brief Title: Feasibility of Using Surplus qFIT Samples to Investigate the Gut Microbiota.
Acronym: FUTURISTIC
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 502
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Gut Microbiota
Keywords: qFIT; Bowel Screening Programme; Gut microbiome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Faecal sample with gut microbiota DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 16 Healthy people: The volunteers will be healthy men and women aged 18 to 65 with a BMI between 18.5 and 30 kg/m2. Volunteers will provide a single stool sample to compare 16S rRNA gene sequencing results for gut microbiota between faeces processed from standard stool sample and those collected by the collection device (EXTEL HEMO AUTO MC Collection Picker) used in the Scottish Bowel Screening Programme.
  Interventions: Other: No intervention
- 100 anonymised qFIT samples: To determine whether our carefully controlled conditions are replicated in the NHS setting, one hundred anonymised qFIT samples will be obtained from Chemical Pathology Aberdeen Royal Infirmary under NHS Grampian Biorepository ethical approval. Extracted DNA will be quantified by Qubit and run on an agarose gel to determine the intact nature of the DNA.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be provided.

SUMMARY:
The Scottish Bowel Screening Programme is an enormous potential research resource; half a million people in Scotland do their bowel screening test each year. If we could obtain meaningful data on the gut microbiota in these individuals, many clinical questions could be answered using nested case-control studies relating gut microbiota profiles to cancer, obesity, cardiovascular and metabolic diseases and Alzheimer's disease. As individuals are screened from age 50 to 74 years, there would also be excellent opportunities for longer-term longitudinal studies.

Since 2017, the bowel screening programme has used qFIT testing for faecal haemoglobin. Patients collect a tiny (2 miligram) sample of their faeces into 2 mililiter of buffer but only approximately 6 microliter is required for testing. The goal of this study is to investigate whether the large number of patients' samples available from the National Bowel Screening Programme could be used in future gut microbiome studies using the leftover faeces in buffer in the qFIT tests.

DETAILED DESCRIPTION:
We aim to test the hypothesis that the 2 mg of faeces suspended in buffer reagent in the qFIT cassette will be sufficient to perform 16S rRNA gene sequencing and will yield comparable results to conventionally collected faecal samples, thus allowing us to study the large number of patients' samples available from the National Bowel Screening Programme in future studies.

If we could demonstrate that the DNA from these faeces yields similar results to that from conventionally collected specimens (e.g. 15-20 ml of faeces collected into a 30 ml stool sample pot), this could allow us to study the large number of patients' samples available from the National Bowel Screening Programme in future studies.

Other studies have investigated the potential for using fresh or frozen residual FIT test buffer instead of intact stool samples to measure faecal microbial features by 16S rRNA gene sequencing, using OC-Auto FIT cartridges (Polymedco Inc) which add 10 mg of faeces to 2 ml of buffer, but buffer stability is lower than for the EXTEL collection picker cartridges (7 days vs 32 days at room temperature; 28 days vs 120 days at 2-8oC).

We hypothesise that the small amount of faeces suspended in buffer reagent in the qFIT cassette will be sufficient to perform 16S rRNA gene sequencing and will yield comparable results to conventionally collected faecal samples.

We shall:

1. determine whether 500 ul of buffer/faeces mix from qFIT collection cassettes will yield sufficient DNA for 16S rRNA gene sequencing or whether 1.5 to 2 ml is required
2. compare 16S rRNA gene sequencing of fresh faeces from 16 human volunteers (processed within 24 hours) using qFIT cassettes and conventional faecal collection methods
3. determine the suitability of faeces collected by qFIT, held in the cassette for durations commensurate with samples handled in the Scottish Bowel Screening Programme, up to 14 days
4. quantify the DNA present in 100 qFIT samples surplus to requirements from symptomatic patients from Aberdeen Royal Infirmary, to determine the proportion of samples with adequate DNA for 16S rRNA gene sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Aged 18 to 65
* BMI 18.5 and 30 kg/m2

Exclusion Criteria:

* A member of Prof Kiltie's lab
* Cconsumed antibiotics within the last 3 months
* Pregnant or breastfeeding
* Cannot drop your samples off at the Rowett Institute
* Have any of the following: History of cardiovascular disease/stroke, diabetes, gastrointestinal disease, autoimmune disorders or cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy people between 18 and 65 years old.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Microbial composition using 16S sequencing. | 5 months
  Comparison of 16S rRNA gene sequencing of fresh faeces processed within 24 hours from 16 human volunteers using qFIT collection cassettes and conventional faecal collection methods.

SECONDARY OUTCOMES:
DNA yield over time, quantified by Qubit | 6 months
  Determination of the suitability of faeces collected by qFIT based on the microbial DNA yield when held in the cassette for durations commensurate with samples handled in the Scottish Bowel Screening Programme. The extracted DNA will also be send for 16S DNA sequencing.
Comparison DNA yield from 16 volunteers with NHS setting | 10 months
  To determine whether our carefully controlled conditions are replicated in the NHS setting, one hundred anonymised qFIT samples, held for 7-14 days post-sample analysis, will be obtained from Chemical Pathology Aberdeen Royal Infirmary under NHS Grampian Biorepository ethical approval. Extracted DNA will be quantified by Qubit (2 ul volume; can detect 0.2 ng to 100 ng) and run on an agarose gel with SYBR Safe fluorescent dye to determine the intact nature of the DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Kiltie, Prof, Principal Investigator — University of Aberdeen
Locations (1):
- Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baxter NT, Koumpouras CC, Rogers MA, Ruffin MT 4th, Schloss PD. DNA from fecal immunochemical test can replace stool for detection of colonic lesions using a microbiota-based model. Microbiome. 2016 Nov 14;4(1):59. doi: 10.1186/s40168-016-0205-y. PMID 27842559
- [Background] Vogtmann E, Chen J, Amir A, Shi J, Abnet CC, Nelson H, Knight R, Chia N, Sinha R. Comparison of Collection Methods for Fecal Samples in Microbiome Studies. Am J Epidemiol. 2017 Jan 15;185(2):115-123. doi: 10.1093/aje/kww177. Epub 2016 Dec 16. PMID 27986704